CLINICAL TRIAL: NCT00904865
Title: Single Port Access Cholecystectomy Versus Standard Laparoscopic Cholecystectomy - Randomized Study
Brief Title: Single Port Access (SPA) Cholecystectomy Versus Standard Laparoscopic Cholecystectomy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Bucher Pascal, MD, University Hospital Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CER-08-145
Record Dates: First submitted 2009-05-19; First posted 2009-05-20 (Estimated); Last update posted 2009-05-20 (Estimated); Status verified 2009-05

CONDITIONS: Symptomatic Gallbladder Stones; Cholecystitis; Biliary Pancreatitis
Keywords: Single port access; Laparoscopy; cholecystectomy; cholangiography; cosmesis
MeSH Terms: conditions — Cholecystitis | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): SPA cholecystectomy
  Interventions: Procedure: SPA cholecystectomy
- 2 (Other): laparoscopic cholecystectomy
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: SPA cholecystectomy — SPA cholecystectomy
  Arms: 1
Procedure: Laparoscopic cholecystectomy — Laparoscopic cholecystectomy
  Arms: 2

SUMMARY:
Background:

Single port access surgery is a rapidly progressing surgical approach which allows performance of standard laparoscopic surgery through a single transparietal port instead of multiple port accesses.

Objective:

Demonstrate the validity of Single port access (SPA) cholecystectomy compared to multiple ports laparoscopic cholecystectomy.

Hypothesis:

SPA cholecystectomy is associated with decreased parietal and body image trauma compare to multiple ports laparoscopic cholecystectomy. SPA cholecystectomy should be associated with better cosmetic results, may improve postoperative recovery due to lower parietal pain. SPA cholecystectomy may also be associated with decreased rate of parietal complications as lower numbers of transparietal port are placed.

Methods:

All patients offered cholecystectomy, either SPA or multiport cholecystectomy, included in the study will have recognized biliary pathology for which formal indication cholecystectomy are recognized internationally.

Surgical technique, either for SPA cholecystectomy or for multiple ports cholecystectomy, will be the same except, that one surgical technique is achieved through a single transparietal port and the other through multiple ports.

Randomization will be performed before surgeries after patients have given their informed consent to the study.

No specific test or cost will be necessitated by the study. Patients will be informed orally and will receive a short study summary, allowing them to give an informed consent.

Endpoints:

* Morbidity
* Body image and Cosmetic results
* Post-operative pain (opioid sparing effect)
* Operative time
* Hospital stay

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years

Exclusion Criteria:

* Contraindication to laparoscopy
* Liver disease
* Cognitive trouble

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Cosmesis, body image and quality of life scale | at 1 month

SECONDARY OUTCOMES:
Post-operative morbidity | at 30 days
Post-operative pain | 10 days
Operative time | day 1

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Bucher, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospital Geneva, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Background] Bucher P, Pugin F, Buchs N, Ostermann S, Charara F, Morel P. Single port access laparoscopic cholecystectomy (with video). World J Surg. 2009 May;33(5):1015-9. doi: 10.1007/s00268-008-9874-4. PMID 19116734
- [Derived] Bucher P, Pugin F, Buchs NC, Ostermann S, Morel P. Randomized clinical trial of laparoendoscopic single-site versus conventional laparoscopic cholecystectomy. Br J Surg. 2011 Dec;98(12):1695-702. doi: 10.1002/bjs.7689. Epub 2011 Sep 30. PMID 21964736
- [Derived] Steinemann DC, Raptis DA, Lurje G, Oberkofler CE, Wyss R, Zehnder A, Lesurtel M, Vonlanthen R, Clavien PA, Breitenstein S. Cosmesis and body image after single-port laparoscopic or conventional laparoscopic cholecystectomy: a multicenter double blinded randomised controlled trial (SPOCC-trial). BMC Surg. 2011 Sep 12;11:24. doi: 10.1186/1471-2482-11-24. PMID 21910897